CLINICAL TRIAL: NCT03135951
Title: Pharmacokinetics of SPI-2012 (Eflapegrastim) in Breast Cancer Patients Receiving Docetaxel and Cyclophosphamide (TC) Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-GCF-301-PK
Record Dates: First submitted 2017-04-20; First posted 2017-05-02 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Breast Cancer; Pharmacokinetics
Keywords: Breast Cancer; Pharmacokinetics; Long-acting Myeloid Growth Factor; Early Stage Breast Cancer; Docetaxel + Cyclophosphamide (TC) Chemotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — eflapegrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SPI-2012 (Experimental): * SPI-2012 (13.2 mg/0.6 mL fixed dose, equivalent to 3.6 mg G-CSF per cycle)
  * Supplied in 1 mL prefilled, single-use syringes for subcutaneous injection
  * Administered on Day 2 of each cycle after TC administration
  Interventions: Drug: SPI-2012

INTERVENTIONS:
Drug: SPI-2012 — Supplied in prefilled, single-use syringes for subcutaneous injection and administered on Day 2 of each cycle.
  Other Names: Rolontis™; Eflapegrastim

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic (PK) profile of a fixed dose of SPI-2012 in patients with early-stage breast cancer receiving docetaxel and cyclophosphamide (TC) chemotherapy, as measured by the serum concentration of SPI-2012 on specific days following drug administration.

DETAILED DESCRIPTION:
This is a Phase 1, single-arm multicenter study to evaluate the PK and safety of SPI-2012 (a long acting myeloid growth factor) in breast cancer patients treated with TC chemotherapy.

Approximately 25 patients will be enrolled.

Each cycle will be 21 days and patients will receive 4 cycles of treatment with 2 additional cycles based on the investigator's discretion. On Day 1 of each cycle, patients will receive TC chemotherapy and on Day 2 of each cycle, patients will receive SPI-2012.

Pharmacokinetics will be evaluated only in Cycles 1 and 3.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, histologically confirmed early-stage breast cancer, defined as operable Stage I to Stage IIIA breast cancer.
* Candidate to receive adjuvant or neoadjuvant TC chemotherapy.
* ANC ≥1.5x10^9/L
* Platelet count ≥100x10^9/L
* Hemoglobin >9 g/dL
* Calculated creatinine clearance >50 mL/min
* Total bilirubin ≤1.5 mg/dL
* AST and ALT ≤2.5xULN
* Alkaline phosphatase ≤2.0xULN
* ECOG ≤2

Exclusion Criteria:

* Active concurrent malignancy (except non melanoma skin cancer or carcinoma in situ of cervix) or life-threatening disease. If history of prior malignancies or contralateral breast cancer, must be disease free for at least 5 years.
* Known sensitivity to E. coli derived products or known sensitivity to any of the products to be administered during dosing.
* Concurrent adjuvant cancer therapy.
* Locally recurrent/metastatic breast cancer.
* Previous exposure to filgrastim, pegfilgrastim, or other G-CSF products in clinical development within 12 months prior to the administration of study drug.
* Active infection, receiving antibiotics or any serious underlying medical condition which would impair the ability of the patient to receive protocol-specified treatment.
* Prior bone marrow or hematopoietic stem cell transplant
* Used any investigational drugs, biologics, or devices within 30 days prior to study treatment or plans to use any of these during the course of the study.
* Prior radiation therapy within 30 days prior to enrollment.
* Major surgery within 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2018-02-19 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Up to 42 days
  PK samples will be collected at predetermined time intervals and Peak Concentration is measured at highest value among all concentrations.
Area under the plasma concentration versus time curve (AUC) | Up to 42 days
  PK samples will be collected at predetermined time intervals. AUC is calculated in the plot of plasma concentration versus time curve

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 6 months
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation patient, temporally associated with the use of a medicinal product or study procedure, whether or not considered related to the medicinal product. A treatment-emergent AE (TEAE) is any AE that occurs from the first dose of study treatment through 35 (±5) days after the date of patient early discontinuation.
Population slope of the relationship between the change from baseline in QTc intervals and plasma concentrations of SPI-2012 | Up to 42 days
  A linear mixed effects modeling approach will be used to quantify the relationship between the plasma concentrations of SPI-2012 and change from baseline in QT intervals (∆QTc). Plasma concentration, intercept, and subject are to be included as random effects.

CONTACTS AND LOCATIONS:
Overall Officials: Shanta Chawla, MD, Study Director — Spectrum Pharmaceuticals, Inc
Locations (1):
- Research Center, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Undecided